CLINICAL TRIAL: NCT02428400
Title: A Phase I/IB Randomized, Double-blind, Placebo Controlled, Dose-finding Study to Evaluate Safety, Tolerability of TG1050 Single/Multiple Doses, and Evaluation of TG1050 Immunologic/Antiviral Activity in Patients With Chronic Hep B Infection
Brief Title: Safety and Tolerability of TG1050: A Dose-finding Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1050.02
Record Dates: First submitted 2015-03-18; First posted 2015-04-28 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TG1050 (Experimental): TG1050 SD cohort, administered SC as a single injection: 9.0 Log [10^9] 10.0 Log [10^10], 11.0 Log [10^11] virus particles
  TG1050 MD cohort, administered SC as 3 once weekly injections:9.0 Log [10^9] 10.0 Log [10^10], 11.0 Log [10^11] virus particles
  TG1050 Part B cohort, dose(s) and schedule to be determined
  Interventions: Biological: TG1050
- Placebo (Placebo Comparator): Placebo SD cohort, administered SC as a single injection: 9.0 Log [10^9] 10.0 Log [10^10], 11.0 Log [10^11] virus particles
  Placebo MD cohort, administered SC as 3 once weekly injections: 9.0 Log [10^9] 10.0 Log [10^10], 11.0 Log [10^11] virus particles
  Placebo Part B cohort, dose(s) and schedule to be determined
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TG1050 — TG1050: adenovirus serotype 5 vector based immunotherapeutic product in adenovirus reference material (ARM) buffer
  Arms: TG1050
Biological: Placebo — Placebo: adenovirus reference material (ARM) buffer
  Arms: Placebo

SUMMARY:
Methodology:

This is a double-blind, randomized, placebo-controlled, multi-cohort Phase 1/1b study in patients that are currently being treated for chronic HBV infection. For all cohorts, patients must be receiving antiviral treatment with either tenofovir disoproxil fumarate (TDF) or entecavir (ENT) for at least two years, and have their HBV infection well-controlled

ELIGIBILITY:
Inclusion Criteria:

* 18 through 65 years of age, inclusive
* Patients must be undetectable for neutralizing antibodies to Adenovirus serotype 5 (Ad5) (PART A ONLY)
* Negative serum β-HCG (for women of childbearing potential only; women of non-childbearing potential are defined as a woman who has been postmenopausal for ≥ 2 years or who had had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure)
* Female patients of childbearing potential must be willing to use double effective methods of contraception (e.g. two of the following: hormonal contraception, condom or occlusive cap, intrauterine device (IUD) or intrauterine system (IUS), male sterilisation, or true abstinence) through 3 months after the last IMP administration; male patients must agree to use a double effective method of contraception (e.g. two of the following: hormonal contraception, condom or occlusive cap, IUD or IUS, male sterilisation, or true abstinence) during heterosexual intercourse with a partner capable of becoming pregnant throughout 3 months after the last IMP administration
* Currently on treatment for HBV monoinfection (any HBV genotypes) for at least 2 years with either the nucleos(t)ide analogue TDF or ENT
* A history of HBV DNA < 20 IU/mL for at least 6 months before entry and HBV DNA < 20 IU/mL at screening.
* HBsAg positive
* HBeAg positive or HBeAg negative patients with HBV infection
* Compensated liver disease; defined as direct or conjugated bilirubin ≤ 1.2 × ULN, PT/INR ≤ 1.2 × ULN, platelets ≥ 150,000/mm3, serum albumin ≥ 3.5 g/L, and no prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)
* ALT ≤ 1.5 x ULN. Due to its biological variability, a re-test of the ALT parameter is allowed if the ALT value at screening does not exceed 10% of the 1.5 x ULN value and all other eligibility criteria are met. In this case, the ALT re-test can be performed no more than one month after the initial ALT screening assay and has to be confirmed within 2 weeks. Values of the two ALT assays re-tests have to be below 1.5 x ULN to include the patient. In case of re-test of the ALT parameter, all hematology and biochemistry parameters will be reassessed in parallel of the second ALT re-test to ensure that they are still matching TG1050.02 eligibility criteria.• Hemoglobin ≥ 10 g/L
* Creatinine clearance > 50mL/min
* Neutrophils ≥ 1,500/mm3
* Signed, written Independent Ethics Committee (IEC)-approved informed consent

Exclusion Criteria:

* Patients with any evidence of hepatocellular carcinoma or any other liver cancer
* Patients with α-fetoprotein > 50 ng/mL
* Patients co-infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis Delta virus (HDV)
* Patients with either a) medical history or evidence of cirrhosis who had any biopsy showing cirrhosis or any approved non-invasive test indicative of cirrhosis as documented in the medical source documents; OR b) either of the following at screening: transient elastography score ≥ 10.5 kPa OR a Fibrotest® Fibrosure® score of ≥ 0.48 and an aspartate aminotransferase platelet ratio Index (APRI) of ≥1. Note: If a biopsy or non-invasive test has never been performed or if a biopsy or non-invasive test has been performed but showed no cirrhosis, then b) must be followed at screening
* Patients with a history of uncontrolled thyroid disease or abnormal thyroid stimulating hormone (TSH) levels at screening (defined as < 0.8 × lower limit of normal [LLN] or > 1.2 × ULN; patients are eligible with abnormal TSH levels if the free triiodothyronine (FT3) and free thyroxine (FT4) are within normal limits)
* Significant concomitant medical disorder including active systemic infection or proven or suspected immunosuppressive disorder
* History of immunodeficiency or autoimmune disease (including autoimmune hepatitis, or preexisting autoimmune or antibody-mediated disease)
* Current or history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, renal, cardiovascular, metabolic, endocrine, neurologic, hematologic illness, major organ transplantation, or any other major medical disorder that, in the judgment of the investigator, would interfere with patient treatment, or preclude patient participation in this study; should be discussed case by case with the Sponsor
* Pregnant or breast-feeding women
* Prior treatment with an experimental gene therapy product or a gene therapy product
* Prior participation in another research protocol involving an investigation medicinal product (IMP) within 4 months prior to TG1050/placebo injection
* History of substance abuse, including alcohol abuse that in the judgment of the investigator would deem the patient as not be suitable for participation in the study
* Patients unable or unwilling to comply with the protocol requirements

All key inclusion and exclusion criteria remain the same for patients in Part A, MD Cohort and in Part B of the study except for the following:

Patients with detectable or undetectable anti-Ad5 neutralizing antibodies are eligible (i.e. regardless of their pre-immunity to Ad5 nAb).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TG1050 administered as single or multiple doses: Overall number of AEs, including SAEs, Grade 3 or 4 AEs, Grade 3 or 4 laboratory abnormalities, and any AE leading to a permanent discontinuation of IMP for any reason. | Week 54
Dosage of TG1050/placebo administration for investigation in Part B of the study will be determined. | Week 54

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (3):
  - Edmonton, Alberta
  - Calgary
  - Montreal
- France (5):
  - Grenoble
  - Lyon
  - Nancy
  - Paris
  - Strasbourg
- Germany (4):
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Mainz